CLINICAL TRIAL: NCT03611907
Title: Prospective Randomized Controlled Trial Comparing Different Needles for Oocyte's Retrieval.
Brief Title: Comparing Two Types of Needle for Oocytes Retrieval
Acronym: NEEDLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1965
Record Dates: First submitted 2018-06-26; First posted 2018-08-02 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Infertility, Female; ART
MeSH Terms: conditions — Infertility, Female | interventions — Oocyte Retrieval

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled clinical trial is designed to highlight differences between Double Lumen Aspiration Needle and Single Lumen Needle commonly used in clinical practice primarly in terms of number of retrieved oocytes per procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SL1(Cook® Single Lumen) (Active Comparator): Oocyte retrieval with only aspiration system
  Interventions: Device: Oocyte retrieval with only aspiration system "SL1(Cook® Single Lumen)"
- DL1 (Cook® EchoTip® Double Lumen) (Active Comparator): Oocyte retrieval with aspiration and flushing system
  Interventions: Device: Oocyte retrieval with aspiration and flushing system "DL1 (Cook® EchoTip® Double Lumen)"

INTERVENTIONS:
Device: Oocyte retrieval with only aspiration system "SL1(Cook® Single Lumen)" — In this intervention a 17-Gauge needle is used to aspirate the follicles
  Arms: SL1(Cook® Single Lumen)
Device: Oocyte retrieval with aspiration and flushing system "DL1 (Cook® EchoTip® Double Lumen)" — In this intervention a 17-Gauge needle is used to aspirate follicle, and consequently a 1 mL flush is injected and aspirated twice for each punctured follicle
  Arms: DL1 (Cook® EchoTip® Double Lumen)

SUMMARY:
In the early stages of assisted reproductive technologies (ART), oocyte retrieval was performed via laparoscopy, a cumbersome and expensive process requiring general anesthesia. Today, transvaginal oocyte retrieval for ART is a routine procedure performed under ultrasound guidance. Double-lumen retrieval needles, which are capable of flushing ovarian follicles, were developed to overcome the possibility of oocyte retention within the ovarian follicles and retrieval collection system. Single lumen needles have been introduced and are routinely used by most groups due to their supposed ability to retrieve the same number of oocytes in a shorter operation time.

DETAILED DESCRIPTION:
After a long period in which Humanitas department used double lumen needles for oocytes retrieval in the last four years the choice of the needle is an operator choice, usually influenced by the number of follicles present at human Chorionic Gonadotropin (hCG) trigger.

This prospective randomized controlled clinical trial is designed to highlight differences between Double Lumen Aspiration Needle and Single Lumen Needle commonly used in Humanitas' clinical practice primarly in terms of number of retrived oocytes per procedure (A). Secondary outcomes are the number of punctured follicles (B), the retrieval rate (%) (A/B), the number of follicles at the last ultrasound performed prior to the ovulation trigger (C), the number of retrieved oocytes / number of follicles at trigger-day (A/C), retrieval procedure time (D), single oocyte retrieval time (D/A), the number of mature oocytes (and MII) and complications rate. Number of transferred embryos, number of frozen embryos and oocytes, clinical pregnancy rate per retrieval and per transfer (considering the number of pregnancies diagnosed by US visualization of one or more gestational sacs or definitive clinical signs of pregnancy per 100 cycles) and total number of clinical pregnancies with fetal heart beat (confirmed by visualization of one or more embryos with heartbeat at early dating ultrasound), are also evaluated. Standard protocols will be used for controlled ovarian hyper stimulation. Trans vaginal ultrasound-guided oocyte retrieval will be performed 36 hours ± 2 after hCG injection with the patient under deep sedation.

One hundred patients per each needle will be enrolled in this trial.

ELIGIBILITY:
Inclusion Criteria:

* IVF/ intracytoplasmatic sperm injection (ICSI) cycles;

Exclusion Criteria:

* Ovarian Endometriomas;
* Severe previous pelvic inflammatory disease with frozen pelvis

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Number of retrieved oocytes per procedure | through study completion, 9 months
  Comparison of the number of retrieved oocytes per procedure among the two arms

SECONDARY OUTCOMES:
Time for single oocyte retrieval (minutes) | through study completion, 9 months
  comparison between the recovery time for single oocyte in days among the two arms
Percentage of MII oocytes retrieved | through study completion, 9 months
  A comparison between the percentage of MII oocytes retrieved among the two arms
Oocyte retrieval percentage per aspirated follicles | through study completion, 9 months
  Comparison between the oocyte retrieval percentage per aspirated follicles among the two arms
number of punctured follicles | through study completion, 9 months
  Comparison of the number of punctured follicles among the two arms
number of follicles at the trigger day | through study completion, 9 months
  Comparison of the number of follicles at the trigger day among the two arms
the number of retrieved oocytes/ number of follicles at the trigger day | through study completion, 9 months
  Comparison of the number of retrieved oocytes/ number of follicles at the trigger day among the two arms
time of the single procedure | through study completion, 9 months
  Comparison of the time of the single procedure among the two arms
Complication rate | through study completion, 9 months
  Comparison of the complication rate among the two arms

CONTACTS AND LOCATIONS:
Locations (1):
- Paolo Emanuele Levi Setti, Rozzano, MI, Italy

REFERENCES:
- [Derived] Ronchetti C, Cirillo F, Immediata V, Gargasole C, Scolaro V, Morenghi E, Albani E, Patrizio P, Levi-Setti PE. A Monocentric Randomized Controlled Clinical Trial to Compare Single- and Double-Lumen Needles in Oocyte Retrieval Procedure in Assisted Reproductive Technologies. Reprod Sci. 2023 Sep;30(9):2866-2875. doi: 10.1007/s43032-023-01232-w. Epub 2023 Apr 17. PMID 37069472